CLINICAL TRIAL: NCT03977571
Title: Multicenter Randomized Trial of Deferred Cytoreductive Nephrectomy in Synchronous Metastatic Renal Cell Carcinoma Receiving Checkpoint Inhibitors: a DaRenCa and NoRenCa Trial Evaluating the Impact of Surgery or No Surgery. The NORDIC-SUN-Trial
Brief Title: Deferred Cytoreductive Nephrectomy in Synchronous Metastatic Renal Cell Carcinoma: The NORDIC-SUN-Trial
Acronym: NORDIC-SUN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Niels Fristrup (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Niels Fristrup, MD PhD, University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NORDIC-SUN
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Kidney Cancer; Renal Cell Carcinoma Metastatic; Synchronous Neoplasm
Keywords: Cytoreduction Surgical Procedures; Nephrectomy; Ipilimumab; Nivolumab; Laboratory biomarker analysis; Gene Expression; Liquid Biopsy
MeSH Terms: conditions — Kidney Neoplasms; Neoplasms, Multiple Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deferred nephrectomy (Experimental): Surgery after induction therapy with IO/IO or a TKI/IO-combination, followed by maintenance therapy with nivolumab or a TKI/IO-combination.
  Interventions: Procedure: Cytoreductive nephrectomy; Other: Tissue sampling
- No surgery (Active Comparator): Induction therapy wih IO/IO or a TKI/IO-combination, followed by maintenance therapy with nivolumab or a TKI/IO-combination.
  Interventions: Other: Tissue sampling

INTERVENTIONS:
Procedure: Cytoreductive nephrectomy — Partial or complete nephrectomy by open, laparoscopic, or robotic approach.
  Arms: Deferred nephrectomy
Other: Tissue sampling — Tumor biopsies, blood, and stool specimens for translational biomarker research will be sampled at baseline and after 3 or 6 months.

SUMMARY:
BACKGROUND: For synchronous metastatic renal cell carcinoma (RCC), surgical resection of the primary tumor in the presence of distant metastases has been the standard of therapy for select patients followed by systemic therapy. In the era of TKIs two randomized trials, CARMENA and SURTIME, have questioned the role and timing of surgery in these patients, results point towards no surgery or a deferred approach.

RATIONALE: The antitumor activity of immune checkpoint blockage (ICB) is more potent than other therapy in mRCC. The deferred cytoreductive nephrectomy approach ensures systemic therapy for all patients, avoid systemic treatment delay, and spare surgery in patients with progressive tumors. Current data only point towards a survival benefit for cytoreductive nephrectomy in intermediate risk patients, but not in poor risk patients

HYPOTHESIS: Deferred cytoreductive nephrectomy after initial nivolumab combined with ipilimumab or a TKI/IO-combination will improve OS in patients with synchronous metastatic RCC and ≤3 IMDC risk features

This is an open, randomized, multicenter comparison trial, designed to evaluate the effect of deferred cytoreductive nephrectomy compared with no surgery following initial nivolumab combined with ipilimumab or a TKI-combination, in mRCC patients with IMDC intermediate and poor risk.

DETAILED DESCRIPTION:
OUTLINE: This is a multicenter trial, patients are stratified according to institution, treatment choice, number of IMDC risk factors, and combined elevated neutrophil-lymphocyte ratio and hyponatremia.

All patients will receive induction checkpoint immunotherapy immediately after inclusion. After 3 months or a total of 4 series of nivolumab combined with ipilimumab or a TKI/IO-combination, the patient will be discussed for resectability at the multidisciplinary meeting (MDT). Whether the patient is eligible for cytoreductive nephrectomy is at the discretion of the urologist at the local MDT. Patients with ≤ 3 IMDC risk factors and deemed suitable for cytoreductive nephrectomy will then undergo randomization. Patients deemed not suitable for surgery or have > 3 IMDC risk features at the 3 month evaluation continue systemic therapy for 3 months, followed by a 2nd evaluation. Patients with ≤ 3 IMDC risk factors and deemed suitable for cytoreductive nephrectomy at 2nd evaluation will then undergo randomization. Patients deemed not suitable for surgery or have > 3 IMDC risk features at the 6 month evaluation continue systemic therapy. Nivolumab may continue until unacceptable toxicity or total treatment length of 2 years from inclusion.

ARM A: Deferred cytoreductive nephrectomy, followed by maintenance nivolumab or a TKI/IO-combination.

ARM B: No surgery, receive maintenance nivolumab or a TKI/IO-combination.

Patients undergo tumor tissue, blood, and stool collection at baseline, 3 and 6 months, for planned translational research.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent obtained prior to any study specific procedures.
2. Patient must be willing and able to comply with the protocol.
3. Age ≥18.
4. Core needle biopsy proven metastatic renal cell carcinoma - all histologic subtypes acceptable.
5. Synchronous metastatic renal cell carcinoma with the primary tumor present in the kidney.
6. Measurable disease as per RECIST v 1.1
7. Patients for which Nivolumab/Ipilimumab or a TKI/IO-combination is considered indicated according to the recommendations by the European Medicines Agency and the national health authorities of participating countries. The prescription of nivolumab/ipilimumab or a TKI/IO-combination in the circumstances of the study is considered as a standard treatment.
8. Females with a negative serum pregnancy test unless childbearing potential can be otherwise excluded (postmenopausal, hysterectomy or oophorectomy) and not lactating.
9. Fertile women of childbearing potential (<2 years after last menstruation) and men must use effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgical sterilization).
10. Karnofsky Performance status ≥70
11. Life expectancy of greater than 4 months.
12. The required laboratory values are as follows:

    * Adequate bone marrow function (Leucocytes > 3.0 x 109/l, platelets > 100 x 109/l, hemoglobin > 6.0 mmol/l or > 10.0 g/dL.)
    * International normalized ratio (INR) ≤ 1.2 x upper limit of normal (ULN)
    * Adequate hepatic function (bilirubin ≤ 1.5 x ULN, ALAT ≤ 2.5 x ULN or ≤ 5 x ULN if liver lesions)
    * Adequate kidney function (eGFR > 35 mL/min)

Exclusion Criteria:

1. Prior systemic treatment for mRCC
2. Other cancer within 3 years (except in situ basal cell carcinoma and localised prostate cancer with undetectable PSA).
3. Major surgical procedure, open surgical biopsy, or significant traumatic injury within 28 days prior to enrollment
4. Clinically significant (i.e active) cardiovascular disease for example cerebrovascular accidents (< 6 months before inclusion), myocardial infarction (< 6 months before inclusion), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure.
5. No symptomatic brain metastasis requiring systemic corticosteroids (> 10 mg daily prednisone equivalent)
6. Recent (within the 30 days prior to inclusion) treatment with another investigational drug or participation in another investigational study.
7. Any active or recent history of a known or suspected autoimmune disease or recent history of a condition that require systemic corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications, excluding inhaled steroids and topical steroids. Subjects with vitiligo or type I diabetes mellitus or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, psoriasis not requiring systemic treatment are permitted to enroll.
8. Known hypersensitivity to monoclonal antibodies.
9. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
10. Any positive test for hepatitis B- or C-Virus indicating acute or chronic infection.
11. Oral or i.v. antibiotics administered 14 days prior to initiation of systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Minimum 3 years follow-up
  Calculated from the date of inclusion, to the date of death of any cause or censored at the date at last follow-up.

SECONDARY OUTCOMES:
Progression free survival | 3 years follow-up
  According to the RECIST v1.1
Time to subsequent systemic therapy | 3 years follow-up
  Calculated from date of inclusion to date of initiation of subsequent therapy or death of any cause or censored at the date of last follow-up
Objective response rate | 3 years follow-up
  According to the RECIST v1.1
Rate of patients meeting randomization criteria | 3 or 6 months
  Compared with baseline values
Fractional percentage of tumor volume (ratio of primary tumor measurement to total sum of target lesions) to survival outcome in deferred cytoreductive nephrectomy patients and no surgery patients | 3 years follow-up
  Compared with baseline values
Number of participants with treatment-related adverse events as by Common Terminology Criteria for Adverse Events version 5.0. | 3 years follow-up
  Evaluation of adverse events
Number of participant with surgical morbidity assessed according to the Clavien-Dindo classification of surgical complications | 3 years follow-up
  Evaluation of surgical morbidity
Tumor infiltrating lymphocytes baseline and after surgery compared with OS, PFS, TST, ORR | 3 year follow-up
  As part of a biomarker analysis
Immune subsets in blood measured by flowcytometry in serial samples compared with OS, PFS, TST, ORR. | 3 year follow-up
  As part of a biomarker analysis
Genetic profile of circulation tumor DNA measured by Next generation sequencing (NGS), compared with OS, PFS, TST, ORR. | 3 year follow-up
  As part of a biomarker analysis
Genetic profile of primary tumor tissue measured by measured by NGS compared with OS, PFS, TST, ORR. | 3 year follow-up
  As part of a biomarker analysis
Profile of gut microbiome measured by NGS compared OS, PFS, TST, ORR. | 3 year follow-up
  As part of a biomarker analysis

CONTACTS AND LOCATIONS:
Overall Officials: Niels Fristrup, MD PhD, Principal Investigator — Department of Oncology, Aarhus University Hospital.
Locations (4):
- Denmark (3):
  - Department of Oncology, Aarhus University Hospital, Aarhus, Central Region of Denmark
  - Department of Oncology, Herlev Hospital, Herlev, Herlev
  - Department of Oncology, Odense University Hospital, Odense
- Department of Urology, Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Iisager L, Ahrenfeldt J, Donskov F, Ljungberg B, Bex A, Lund L, Lyskjaer I, Fristrup N. Multicenter randomized trial of deferred cytoreductive nephrectomy in synchronous metastatic renal cell carcinoma receiving checkpoint inhibitors: the NORDIC-SUN-Trial. BMC Cancer. 2024 Feb 24;24(1):260. doi: 10.1186/s12885-024-11987-3. PMID 38402173
- [Derived] Kuusk T, Abu-Ghanem Y, Mumtaz F, Powles T, Bex A. Perioperative therapy in renal cancer in the era of immune checkpoint inhibitor therapy. Curr Opin Urol. 2021 May 1;31(3):262-269. doi: 10.1097/MOU.0000000000000868. PMID 33742979